CLINICAL TRIAL: NCT03592940
Title: Association Between Mediterranean Diet and Neuroendocrine Tumours.
Brief Title: The Management of Neuroendocrine Tumours: A Nutritional Viewpoint.
Acronym: NetNutr
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Prof. Silvia Savastano, Associate Professor, Federico II University
Other Study IDs: 201/17
Record Dates: First submitted 2018-07-10; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Mediterranean Diet; Neuroendocrine Tumours (NETs)
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Diet, Mediterranean

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Mediterranean diet — We aim to determine the effects of the traditional Mediterranean Diet on neuroendocrine tumours

SUMMARY:
Nutritional status in patients with neuroendocrine tumours (NETs), especially of gastroenteropancreatic origin, can be deeply affected by excessive production of gastrointestinal hormones, peptides, and amines, which can lead to malabsorption, diarrhoea, steatorrhea, and altered gastrointestinal motility. Besides, the surgical and/or medical management of NETs can lead to alteration of gastrointestinal secretory, motor, and absorptive functions, with both dietary and nutritional consequences. Indeed, disease-related malnutrition is a frequently encountered yet both underrecognized and understudied clinical phenomenon in patients with NETs, with substantial prognostic and socioeconomic consequences. Most of these conditions can be alleviated by a tailored nutritional approach, also with the aim of improving the efficacy of cancer treatments. In this setting, skilled nutritionists can play a fundamental role in the multidisciplinary health care team in NETs management and their presence should be recommended.

ELIGIBILITY:
Inclusion Criteria:

* patients with neuroendocrine tumours (NETs)

Exclusion Criteria:

* age>65 years
* < BMI 19 kg/m2
* vegetarians

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: One hundred patients with neuroendocrine tumours (NETs) were consecutively enrolled (aged 18-60 years) in this cross-sectional observational study. Anthropometric measures were evaluated. A validated 14-item questionnaire PREDIMED (PREvención con DIeta MEDiterránea) was used for the assessment of adherence to the MD. Dietary data were collected by a 7-day food records.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Adherence to Mediterranean Diet by Predimed Questionnaire | December 2017 to June 2018
  Validated 14-item tool of adherence to the Mediterranean diet, with three categories of adherence (≤5, low adherence, 6-9, average adherence and ≥10 points, high adherence)

SECONDARY OUTCOMES:
Body composition | December 2017 to June 2018
  BIA was performed using a BIA phase-sensitive system by experienced observers (an 800-µA current at a frequency single-frequency of 50 kHz BIA 101 RJL, Akern Bioresearch, Florence, Italy)

CONTACTS AND LOCATIONS:
Locations (1):
- Silvia Savastano, Naples, Italy

IPD SHARING:
Plan to Share IPD: No